CLINICAL TRIAL: NCT00716534
Title: A Phase 2 Randomized, Placebo-Controlled, Double-Blind Study of Carboplatin/Paclitaxel in Combination With ABT-869 Versus Carboplatin/Paclitaxel Alone in Subjects With Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC) as First-Line Treatment
Brief Title: Study of Carboplatin/Paclitaxel in Combination With ABT-869 in Subjects With Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M10-301; 2007-007107-32 (EudraCT Number)
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Advanced or Metastatic Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — linifanib; Carboplatin; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- A (Experimental): 12.5 mg ABT-869 + Carboplatin/Paclitaxel
  Interventions: Drug: ABT-869; Drug: Carboplatin; Drug: Paclitaxel
- B (Experimental): 7.5 mg ABT-869 + Carboplatin/Paclitaxel
  Interventions: Drug: ABT-869; Drug: Carboplatin; Drug: Paclitaxel
- C (Placebo Comparator): Placebo (7.5 mg or 12.5 mg) + Carboplatin/Paclitaxel
  Interventions: Drug: Placebo for ABT-869; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: ABT-869 — 12.5 mg ABT-869
  Arms: A
Drug: Placebo for ABT-869 — Placebo Comparator (12.5 mg or 7.5 mg)
  Other Names: Placebo
  Arms: C
Drug: ABT-869 — 7.5 mg ABT-869
  Arms: B
Drug: Carboplatin — Carboplatin (AUC 6 mg/mL/min)
Drug: Paclitaxel — Paclitaxel (200 mg/m2)

SUMMARY:
This study is designed to determine the clinical efficacy and toxicity of ABT-869 in combination with carboplatin and paclitaxel in the treatment of subjects with advanced or metastatic NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age.
* Subject must have cytologically or histologically confirmed non-squamous NSCLC
* Subject must have recurrent or advanced (Stage IIIb with pleural or pericardial effusion) or metastatic (Stage IV) disease that is not amenable to surgical resection or radiation with curative intent.
* Subject has measurable disease, defined as at least 1 unidimensional measurable lesion on a computed tomography (CT) scan as defined by RECIST (for subjects in the randomized portion only).
* Subject has an ECOG Performance Score of 0-1.
* Willing to take adequate measures to prevent pregnancy.

Exclusion Criteria:

* The subject has NSCLC with a predominant squamous cell histology
* Subject has hypersensitivity to paclitaxel.
* Subject has received any anti-cancer therapy for treatment of NSCLC.
* Subject has received radiation therapy within 21 days of Study Day 1.
* Subject has had major surgery within 21 days.
* Subject has untreated brain or meningeal metastases.
* Subject is receiving therapeutic anticoagulation therapy.
* Subject has a central thoracic tumor lesion as defined by location within the hilar structures.
* Subject has proteinuria CTC Grade > 1 at baseline.
* Subject has a history of, or currently exhibits clinically significant cancer related events of bleeding.
* The subject currently exhibits symptomatic or persistent, uncontrolled hypertension defined as diastolic blood pressure (BP) > 90 mm Hg or systolic BP > 140 mm Hg.
* The subject has a history of myocardial infarction, stroke or Transient Ischemic Attack (TIA) within 6 months of Study Day 1.
* The subject has a documented left ventricular (LV) ejection fraction < 50%.
* The subject has known autoimmune disease with renal involvement (i.e., lupus).
* The subject is receiving combination anti-retroviral therapy for HIV.
* The subject has clinically significant uncontrolled condition(s).
* The subject has a history of another active cancer within the past 5 years.
* The subject has active ulcerative colitis, Crohn's disease, celiac disease or any other conditions that interfere with absorption.
* The subject has a medical condition, which in the opinion of the study investigator places them at an unacceptably high risk for toxicities.
* The subject is pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2008-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Disease Progression

SECONDARY OUTCOMES:
Overall survival, best response rate, time to tumor progression, objective response rate, best percent change in tumor size, duration of response | Disease Progression
Survival Rate | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Justin L. Ricker, MD, Study Director — AbbVie
Locations (37):
- United States (13):
  - Site Reference ID/Investigator# 15850, Chandler, Arizona
  - Site Reference ID/Investigator# 15846, Peoria, Arizona
  - Site Reference ID/Investigator# 15841, Miami, Florida
  - Site Reference ID/Investigator# 7179, Atlanta, Georgia
  - Site Reference ID/Investigator# 15851, Lansing, Michigan
  - Site Reference ID/Investigator# 15844, Lebanon, New Hampshire
  - Site Reference ID/Investigator# 22443, Hackensack, New Jersey
  - Site Reference ID/Investigator# 15848, Greensboro, North Carolina
  - Site Reference ID/Investigator# 22444, Canton, Ohio
  - Site Reference ID/Investigator# 15847, Cleveland, Ohio
  - Site Reference ID/Investigator# 26842, Hershey, Pennsylvania
  - Site Reference ID/Investigator# 13101, Philadelphia, Pennsylvania
  - Site Reference ID/Investigator# 24122, Philadelphia, Pennsylvania
- Australia (4):
  - Site Reference ID/Investigator# 19042, Bedford Park
  - Site Reference ID/Investigator# 23682, Cairns
  - Site Reference ID/Investigator# 21862, Lismore
  - Site Reference ID/Investigator# 19043, Woodville South
- Brazil (7):
  - Site Reference ID/Investigator# 17703, Jaú
  - Site Reference ID/Investigator# 23522, Porto Alegre
  - Site Reference ID/Investigator# 15601, Porto Alegre
  - Site Reference ID/Investigator# 17704, Rio de Janeiro
  - Site Reference ID/Investigator# 22684, Santo André
  - Site Reference ID/Investigator# 17702, São Paulo
  - Site Reference ID/Investigator# 23582, São Paulo
- Czechia (5):
  - Site Reference ID/Investigator# 18964, Kyjov
  - Site Reference ID/Investigator# 22504, Náchod
  - Site Reference ID/Investigator# 18963, Olomouc
  - Site Reference ID/Investigator# 18962, Prague
  - Site Reference ID/Investigator# 19022, Pribram V
- Russia (7):
  - Site Reference ID/Investigator# 38003, Kazan'
  - Site Reference ID/Investigator# 38260, Kirov
  - Site Reference ID/Investigator# 18064, Moscow
  - Site Reference ID/Investigator# 18065, Moscow
  - Site Reference ID/Investigator# 23312, Moscow
  - Site Reference ID/Investigator# 18066, Moscow
  - Site Reference ID/Investigator# 23562, Saint Petersburg
- Site Reference ID/Investigator# 18961, Singapore, Singapore

REFERENCES:
- [Derived] Ramalingam SS, Shtivelband M, Soo RA, Barrios CH, Makhson A, Segalla JG, Pittman KB, Kolman P, Pereira JR, Srkalovic G, Belani CP, Axelrod R, Owonikoko TK, Qin Q, Qian J, McKeegan EM, Devanarayan V, McKee MD, Ricker JL, Carlson DM, Gorbunova VA. Randomized phase II study of carboplatin and paclitaxel with either linifanib or placebo for advanced nonsquamous non-small-cell lung cancer. J Clin Oncol. 2015 Feb 10;33(5):433-41. doi: 10.1200/JCO.2014.55.7173. Epub 2015 Jan 5. PMID 25559798